CLINICAL TRIAL: NCT05699499
Title: Analysis of Impact of KeryFlex on Quality of Life for Retronychia or Lichen Planus Adult Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-04024687
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Lichen Planus of Nail
Keywords: Retronychia; KeryFlex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KeryFlex (Experimental): Patients 18 years and older presenting with retronychia and/or lichens planus of the toenails and/or fingernails to the Weill Cornell Medicine, Department of Dermatology, specialized nail clinic.
  Interventions: Other: KeryFlex

INTERVENTIONS:
Other: KeryFlex — KeryFlex is a painless, in-office cosmetic application of artificial nails which improves the appearance of nails damaged by various nail disorders. The composite resin creates a flexible, nonporous nail that allows the remaining natural nail to grow. KeryFlex is a three-step procedure that takes 10 to 15 minutes for a typical nail. At least 15% of the existing nail must be present for the resin application. The material used in KeryFlex is approved as a cosmetic by the FDA.

SUMMARY:
The purpose of this study is to assess the overall effect of KeryFlex study intervention on quality of life and functionality for patients with retronychia or nail lichen planus.

DETAILED DESCRIPTION:
Retronychia is the growth of the proximal nail plate into the proximal nail fold which was first described in 1999 by De Berker and Rendall. The disorder is common and most frequently affects women (~82%); the estimated average age is 39 years. The unilateral hallux is the most commonly diagnosed site, though nails of the hand (especially thumb and index finger) may also be affected. Common triggers of retronychia include minor trauma (e.g., wearing poorly fitting shoes, jogging,) and systemic illness (e.g., arthritis, thrombophlebitis), which cause disruption of the longitudinal nail bed growth and ultimately lead to the new plate growing vertically into the proximal nail fold. The most frequent cause is trauma. Clinical symptoms include pain, inflammation of the proximal nail fold, granulation tissue under the proximal nail fold, and changes in the proximal nail plate such as thickening or yellowing. Diagnosis is confirmed by clinical presentation and ultrasound. Treatment is particularly challenging. Topical corticosteroids have been used with favorable results; however, recurrences are frequent. Complete nail avulsion is used for severe and/or recalcitrant cases, but this is also associated with frequent relapse rates.

Lichen planus is a chronic inflammatory dermatosis involving mucocutaneous surfaces, scalp, and nails. Nail involvement is observed in around 10% of patient and typically affects the fingernails more than toenails. Nail lichen planus can cause extensive scarring and nail loss. Permanent dystrophy in the forms of anonychia and dorsal pterygium has both functional and psychological consequences. Diagnosis is typically clinical, but a punch biopsy of the nail matrix or nail bed may be utilized if a diagnosis is questionable. There is no evidence-based management for nail lichen planus to date, though expert consensus recommends intralesional steroid injections or systemic corticosteroids as first-line treatment. Outcomes are inconsistent with steroid treatment.

KeryFlex nail is defined as a cosmetic by the Food and Drug Administration (FDA). KeryFlex is a painless, in-office aesthetic application of acrylic nails which improves the appearance of nails damaged by various nail disorders. The composite resin creates a flexible, nonporous nail that allows the remaining natural nail to grow. KeryFlex is composed of a resin material which is applied on the affected nails following the next steps: debridement of the nail, application of bond, application of the resin in the desired color, shape, and size, and curing of the resin by an ultraviolet light. The typical interval between KeryFlex applications is 6 to 8 weeks.

Application of an artificial resin nail to the affected digit may help counter burdensome effects of retronychia or nail lichen planus, including impaired social interactions and loss of functionality. There are no other options for symptom management of retronychia or nail lichen planus in the literature to our knowledge. Attachment of an artificial nail to the newly growing nail may also prevent distal embedding caused by dorsal expansion of the distal pulp, a possible complication of the loss of counterpressure induced by the loss of the nail plate after total nail avulsion.6 Nail resin will be applied as part of the study. Importantly, patients with retronychia very often report that their nail does not grow as quickly as the non-affected ones. Therefore, Keryflex application may be particularly useful if these patients, considering that they would not need to replace the Keryflex as often.

KeryFlex, Pod-Advance, Inc. will provide necessary equipment, but it does not pay Weill Cornell Medicine to conduct this study.

At the screening visit, potential participants will be screened by inclusion and exclusion criteria. History will be obtained including review of medications. Nail clipping sample for histopathology will be taken to rule out onychomycosis if a diagnosis of retronychia is unclear.

Patients will be consented and at baseline visit, during which patients will also be asked to take a quality of life survey to assess baseline impact of retronychia on quality of life. Pre-treatment photographs of patient toenails will be taken. KeryFlex will then be applied to patients' affected nails.

Patients will come to clinic eight weeks after baseline visit, at which point patients will be asked to take a repeat quality of life and satisfaction survey. Post-treatment photographs of patient resin nails will be taken. KeryFlex will then be removed, and photographs post-removal will be taken. The typical interval between KeryFlex application is 6 to 8 weeks.

At two-month follow up visit after KeryFlex treatment, patients will be asked to take a repeat quality of life and satisfaction survey. Post-treatment photographs of patient toenails will be taken. KeryFlex resin will be removed, and photographs post-removal will be taken.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of retronychia or nail lichen planus
* Able to understand and voluntarily sign an informed consent form
* 18-95 years old at time of consent
* Able to adhere to the study visit schedule and other protocol requirements

Exclusion criteria:

* Unable to provide written informed consent for any reason
* Diagnosis of peripheral vascular disease, arterial insufficiency, peripheral neuropathy, suspicious pigmented lesions on the nail or in-grown nails
* Sensitive or allergic to any KeryFlex ingredients
* Unable to abstain from using nail polishes, nail gels, or any other nail products 2 days prior to KeryFlex procedure and during the study period
* Pregnant, planning pregnancy, or nursing

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Change in social domain of quality of life, as measured by social domain scale | Baseline; Week 8
  A three-item social domain scale
  Total possible low score in quality of life, social domain: 0 (0=worst quality of life, social domain) Total possible high score in quality of life, social domain: 100 (100=best quality of life, social domain)
Change in emotional domain of quality of life, as measured by emotional domain scale | Baseline; Week 8
  A seven-item emotional domain scale
  Total possible low score in quality of life, emotional domain: 0 (0=worst quality of life, emotional domain) Total possible high score in quality of life, emotional domain: 100 (100=best quality of life, emotional domain)
Change in symptoms domain of quality of life, as measured by symptoms domain scale | Baseline; Week 8
  A three-item symptoms domain scale
  Total possible low score in quality of life, symptoms domain: 0 (0=worst quality of life, symptoms domain) Total possible high score in quality of life, symptoms domain: 100 (100=best quality of life, symptoms domain)

CONTACTS AND LOCATIONS:
Overall Officials: Shari R Lipner, MD PhD, Principal Investigator — Weill Cornell Dermatology
Locations (1):
- Weill Cornell Dermatology, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ventura F, Correia O, Duarte AF, Barros AM, Haneke E. "Retronychia--clinical and pathophysiological aspects". J Eur Acad Dermatol Venereol. 2016 Jan;30(1):16-9. doi: 10.1111/jdv.13342. Epub 2015 Oct 5. PMID 26435476
- [Background] Gerard E, Prevezas C, Doutre MS, Beylot-Barry M, Cogrel O. Risk factors, clinical variants and therapeutic outcome of retronychia: a retrospective study of 18 patients. Eur J Dermatol. 2016 Aug 1;26(4):377-81. doi: 10.1684/ejd.2016.2774. PMID 27122126
- [Background] Maddy AJ, Tosti A. What's New in Nail Disorders. Dermatol Clin. 2019 Apr;37(2):143-147. doi: 10.1016/j.det.2018.12.004. Epub 2019 Feb 14. PMID 30850036
- [Background] Weston G, Payette M. Update on lichen planus and its clinical variants. Int J Womens Dermatol. 2015 Sep 16;1(3):140-149. doi: 10.1016/j.ijwd.2015.04.001. eCollection 2015 Aug. PMID 28491978
- [Background] Lim SS, Chamberlain A, Hur K, Ohn J, Han B, Mar V, Mun JH. Dermoscopic Evaluation of Inflammatory Nail Disorders and Their Mimics. Acta Derm Venereol. 2021 Sep 15;101(9):adv00548. doi: 10.2340/00015555-3917. PMID 34490472
- [Background] Wechsuruk P, Bunyaratavej S, Kiratiwongwan R, Suphatsathienkul P, Wongdama S, Leeyaphan C. Clinical features and treatment outcomes of nail lichen planus: A retrospective study. JAAD Case Rep. 2021 Sep 22;17:43-48. doi: 10.1016/j.jdcr.2021.09.015. eCollection 2021 Nov. No abstract available. PMID 34703863
- [Background] Goettmann S, Zaraa I, Moulonguet I. Nail lichen planus: epidemiological, clinical, pathological, therapeutic and prognosis study of 67 cases. J Eur Acad Dermatol Venereol. 2012 Oct;26(10):1304-9. doi: 10.1111/j.1468-3083.2011.04288.x. Epub 2011 Nov 3. PMID 22049906
- [Background] Iorizzo M, Tosti A, Starace M, Baran R, Daniel CR 3rd, Di Chiacchio N, Goettmann S, Grover C, Haneke E, Lipner SR, Rich P, Richert B, Rigopoulos D, Rubin AI, Zaiac M, Piraccini BM. Isolated nail lichen planus: An expert consensus on treatment of the classical form. J Am Acad Dermatol. 2020 Dec;83(6):1717-1723. doi: 10.1016/j.jaad.2020.02.056. Epub 2020 Feb 26. PMID 32112995
- [Background] Mello CDBF, Souza MDRE, Noriega LF, Chiacchio ND. Retronychia. An Bras Dermatol. 2018 Sep-Oct;93(5):707-711. doi: 10.1590/abd1806-4841.20187908. PMID 30156621